CLINICAL TRIAL: NCT05335083
Title: The Impact of CPAP on Glucose Metabolism in Moderate-Severe Obstructive Sleep Apnoea Patients Without Diabetes - An Observational Study
Brief Title: CPAP and Glucose Metabolism in Non-Diabetic OSA Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021/ETH12082
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Obstructive Sleep Apnea; Pre-diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP off condition (No Intervention): Participants will be monitored for a two-week period prior to commencing CPAP.
- CPAP on condition (Experimental): Participants will be monitored for a two-week period at least four weeks following commencement of CPAP.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — A positive CPAP intervention
  Arms: CPAP on condition

SUMMARY:
The purpose of the current study is to investigate whether alleviation of OSA by CPAP positively impacts glucose metabolism in non-diabetic patients.

DETAILED DESCRIPTION:
Glucose metabolism in patients newly diagnosed with moderate-severe OSA and without diabetes will be monitored for two weeks prior to commencement of CPAP using a CGM. They will consume a 75g oral glucose drink fasted on waking twice during the two-week monitoring period, having consumed a standardised meal the evening prior. After establishing CPAP use for at least four weeks they will undergo the same protocol as for the observation period prior to commencing CPAP. Glucose metabolism will be monitored using an interstitial (skin based) glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Community dwelling adult males and females aged 18-65 years
2. Polysomnography confirmed moderate to severe OSA with apnea hypopnea index (AHI) ≥15/hr within the past 60 months
3. Able to give written informed consent
4. Proficient in English

6. Diagnosed non-diabetic as defined by the American Diabetes Association as any of the following recent (<3 months) findings:

1. Fasting glucose with a BGL <7.0 mmol/L
2. Glucose tolerance with a 2-hour BGL of < 11.1 mmol/L after a formal 75g Oral Glucose Tolerance Test (OGTT)
3. HbA1C of ≤ 6.5% 7. Possession or regular access to a mobile telephone with capability to download and run the Withings Sleep Anlayser App.

Exclusion Criteria:

1. Clinically significant co-morbidity (e.g. myocardial infarction, congestive heart failure, stroke, arrythmia, chronic kidney or liver disease, epilepsy, head injury)
2. Severe mental health disorders (e.g. current major depressive disorder, schizophrenia, bipolar disorder) that in the opinion of the investigator is not adequately treated or will significantly affect their participation in the study.
3. Regular (>2 times per month) use of sleep-affecting medication (e.g. benzodiazepines, opioids, antidepressants)
4. Regular night shift work or travel overseas within the last 2 weeks
5. Sleep physician has advised against CPAP withdrawal
6. Pregnancy
7. Active smoking or routine alcohol use (more than 2 standard drinks a day) or excessive caffeine intake (>300 mg a day) or recent (in the past month) use of illicit drugs
8. Current or previous diagnosis of diabetes mellitus (previous gestational diabetes mellitus not excluded)
9. Current or recent (<3 months) use of hypoglycaemic agents
10. Undergoing a weight loss programme
11. Contraindications for use of the FreeStyle Libre Pro Sensor. E.g. Known hypersensitivity to skin adhesives such as those used to attach the sensor to the arm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Mean 24 hour glucose difference between the CPAP on and CPAP off conditions | 2 weeks
  Average 24 hour glucose difference between CPAP on and CPAP off conditions

SECONDARY OUTCOMES:
Mean daytime glucose difference between the CPAP on and CPAP off conditions | 2 weeks
  Mean Daytime (6:00 AM - 10:00 PM) glucose difference between the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Mean night time glucose | 2 weeks
  Mean Night-time (10:00 PM - 6:00 AM) glucose difference between the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Glucose tolerance | 2 weeks
  Difference in glucose tolerance as measured by peak 2-hour post 75g glucose load administered twice during each two-week observation period using a CGM
Coefficient of Variation | 2 Weeks
  Percentage CV intraday (i.e. within 24h) and interday (i.e. over multiple days) between the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
SD of Mean Glucose | 2 Weeks
  SD of Mean Glucose (daily) during the CPAP on and CPAP off conditions during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Time in Range (TIR) | 2 Weeks
  Percentage of TIR (3.9-10.0 mmol/L) (hours and minutes) during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Time Below Range (TBR) | 2 Weeks
  Percentage of TBR (3.9 mmol/L including readings of <3 .0 mmol/L) during the the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Time below Range <3.0 mmol/L | 2 Weeks
  Percentage of TBR <3.0 mmol/L (hours and minutes) during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Time Above Range (TAR) | 2 Weeks
  Percentage of TAR (>10.0 mmol/L, including readings >13.9 mmol/L) (hours and minutes) during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Time Above Range >13.9 mmol/L | 2 Weeks
  Percentage of TAR >13.9 mmol/L (hours and minutes) during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Time in Tight Range (TITR) | 2 Weeks
  Percentage of TITR (3.9-7.8 mmol/L) (hours and minutes) during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Change in Glucose Management Indicator | 2 Weeks
  Absolute main change in mmol/L or percentage during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Extended hypoglycaemic event rate | 2 Weeks
  Number of events with sensor glucose <3.9 mmol/L lasting at least 120 min, event ends when glucose returns to at least 3.9 mmol/L for at least 15 minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Extended hyperglycaemic event | 2 Weeks
  Number of events with sensor glucose >13.9 mmol/L lasting at least 120 min; event ends when glucose returns to 10 mmol/L or less for at least 15 minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TIR >70% | 2 Weeks
  Proportion of participants with TIR 3.9-10.0 mmol/L for >70% of the day during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TIR improvement at least 5% | 2 Weeks
  Proportion of participants with TIR 3.9-10.0 mmol/L with at least a 5% improvement from baseline during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TIR improvement at least 10% | 2 Weeks
  Proportion of participants with TIR 3.9-10.0 mmol/L with at least a 10% improvement from baseline during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TBR <3.9 mmol/L <4% | 2 Weeks
  Proportion of participants with TBR <3.9 mmol/L for <4% of each day during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TBR <3.0 mmol/L <1% | 2 Weeks
  Proportion of participants with TBR <3.0 mmol/L for <1% of each day during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TAR >10.0 mmol/L >25% | 2 Weeks
  Proportion of participants with a TAR >10.0 mmol/L for <25% of each day during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TAR >13.9 mmol/L <5% | 2 Weeks
  Proportion of participants with TAR >13.9 mmol/L for <5% of each day during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Hypoglycaemia | 2 Weeks
  Number of times CGM sensor values are <3.9 mmol/L (including readings of <3.0 mmol/L) for at least 15 consecutive minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods. The event ends when there is at least 15 consecutive minutes with a CGM sensor value at least 3.9 mmol/L.
Hypoglycaemia Alert Value (Level 1) | 2 Weeks
  Number of times CGM sensor values are 3.0-3.9 mmol/L for at least 15 consecutive minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods. The event ends when there is at least 15 consecutive minutes with a CGM sensor value at least 3.9 mmol/L.
Clinically Significant Hypoglycaemia (Level 2) | 2 Weeks
  Number of times CGM sensor values are <3.0 mmol/L for at least 15 consecutive minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods. The event ends when there is at least 15 consecutive minutes with a CGM sensor value at least 3.0 mmol/L.
Extended Hypoglycaemia | 2 Weeks
  Number of times CGM sensor values are <3.9 mmol/L for at least 120 consecutive minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
High Glucose Level (Level 1) | 2 Weeks
  Number of times CGM sensor values are 10.1-13.9 mmol/L for at least 15 consecutive minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods. The event ends when there is at least 15 consecutive minutes with a CGM sensor value at or below 10 mmol/L.
Very High Glucose (Level 2) | 2 Weeks
  Number of times CGM sensor values are >13.9 mmol/L for at least 15 consecutive minutes during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods. The event ends when there is at least 15 consecutive minutes with a CGM sensor value at or below 13.9 mmol/L.
Extended Hyperglycaemia | 2 Weeks
  Number of times CGM sensor values are >13.9 mmol/L for at least 90 consecutive minutes within a 120-minute period during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.

OTHER OUTCOMES:
TIR Improvement >10% and <0.5% increase in TBR <3.0 mmol/L | 2 Weeks
  Proportion of participants with >10% improvement in percentage of TIR 3.9-10.0 mmol/L without an increase in the TBR <3.0 mmol/L of >0.5% during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
Mean Glucose <8.6 mmol/L and <1% TBR <3.0 mmol/L | 2 Weeks
  Proportion of participants with Mean Glucose <8.6 mmol/L and < 1% TBR <3.0 mmol/L during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TIR >70% and <1% TBR <3.9 mmol/L | 2 Weeks
  Proportion of participants with >70% TIR 3.9-10.0mmol/L and <4% TBR <3.9 mmol/L during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.
TIR >70% and < 1% TBR <3.0 mmol/L | 2 Weeks
  Proportion of participants with >70% TIR 3.9-10.0 mmol/L and <1% TBR <3.0 mmol/L during the CPAP on and CPAP off conditions as measured by the FreeStyle Libre Pro sensor during the 2-week intervention periods.

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Phillips, PhD, Principal Investigator — Woolcock Institute of Medical Research
Locations (2):
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Woolcock Institute of Medical Research, Macquarie Park, New South Wales

IPD SHARING:
Plan to Share IPD: No
All data will be deidentified using a unique study ID.